CLINICAL TRIAL: NCT06734221
Title: STAR-PAK Study: Evaluating the Safety and Efficacy of PAK® (Paclitaxel Coated Balloon) in Treating Atherosclerotic Femoro-Popliteal Lesions
Acronym: STAR-PAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-BAL-0001
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Popliteal Artery Stenosis Above the Knee; Peripheral Artery Disease; Superficial Femoral Artery Stenosis
Keywords: Peripheral Artery Disease; Drug Coated Balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PAK DCB catheter (Experimental): Peripheral revascularization procedure using a PAK DCB catheter covered with paclitaxel.
  Interventions: Device: Paclitaxel Coated Peripheral Angioplasty Balloon Catheter

INTERVENTIONS:
Device: Paclitaxel Coated Peripheral Angioplasty Balloon Catheter — Paclitaxel coated peripheral angioplasty balloon catheters are catheters of "over the wire" (OTW) type. Distal part of the catheter consists of two channels. External channel is used for inflating the balloon, and internal channel is the guide wire. Catheter has two markers enabling precise determination of balloon position in the vessel. The balloon is covered with a coating POLIGRADE® and drug paclitaxel an amount to 2.5 µg/mm2 , which is eluting during balloon inflation. Paclitaxel belongs to alkaloids group from taxanes group. It is cytostatic and it inhibits the cell cycle in G2/M phase. By inhibiting division of cells and their migration, paclitaxel allows for limiting restenosis phenomenon. Paclitaxel selectively inhibits smooth myocytes proliferation, while the endothelium cells show higher resistance to its action. In addition, paclitaxel restricts inflammatory conditions in walls of the arteries after balloon angioplasty.
  Other Names: PAK®

SUMMARY:
The primary objective of the study is to evaluate the performance and the safety of the PAK® DCB Catheter in the treatment of de novo and restenotic atherosclerotic lesions in the superficial femoral and/or popliteal arteries (SFA/PA) of patients with symptomatic peripheral artery disease (PAD).

The study enrolls patients who have been diagnosed with peripheral artery disease with stenosis of the superficial femoral or popliteal artery and are qualified for endovascular revascularization.

Lower extremity peripheral artery disease may be asymptomatic or may be accompanied by clinical symptoms due to restricted blood flow to the lower extremities.

The management of a patient diagnosed with peripheral arteriosclerosis is primarily aimed at reducing symptoms of limb ischemia and improving blood supply to the limb, as well as seeking to halt the progression of the disease.

Treatment of lower extremity atherosclerosis with percutaneous methods is a well-known minimally invasive and recommended treatment for lower extremity ischemia.

A maximum of 120 patients will be included in the study. All patients included in the study will receive treatment with the investigational device.

The study will use the PAK balloon catheter, which is CE certified and approved for the treatment of patients with peripheral vascular disease. That is, it is also used as standard outside the study. The test procedure with the study device is in accordance with its registration and instructions for use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Written informed consent of the patient to participate in the study.
3. Symptoms of lower limb ischemia defined by Rutherford classification from 2 to 4.
4. At least one de novo or restenotic lesion, in SFA and/or PA defined as a lesion with a proximal origin >10mm from SFA origin and a distal end above the knee joint (at least 3 cm above bottom of the femur- P1).
5. Target Lesion >60% stenosis in the SFA or PA (based on angio-CT and/or confirmed in angiography).
6. Target Lesion <150 mm that consists of no more than two adjacent lesions ≤ 25mm apart and is able to be completely covered with inflation of single investigated PAK DCB (with minimum of >5mm proximal and distal margin.

   Note: Adjacent or tandem lesions must be treated as a single lesion.
7. Reference Vessel Diameter (RVD) between 4.0 and 8.0mm and within treatment range of PAK® DCB to be used 1:1 at the target lesion.
8. Angiographic evidence of distal run-off demonstrated by at least one patent tibial vessel without evidence of significant ≥50% angiographic stenosis from origin to ankle.
9. In-flow vessel (both iliac and femoral) without significant ≥50% angiographic stenosis or successful treatment (≤30% residual stenosis with no complications) of a diseased in-flow vessel at least 30 days prior to the index procedure.

Note: treatment of contralateral iliac arteries is allowed.

Exclusion Criteria:

1. Life expectancy less than 2 years.
2. Suspected or detected malignancy without completed treatment (not considered cured).
3. Planned surgical or interventional procedures within 30 days after the study procedure.
4. Known impaired renal function with GFR ≤30 mL/min per 1.73 m2 and/or elevated serum creatinine > 2.5mg/dL or on dialysis.
5. Active inflammatory process at the site of the planned puncture.
6. Acute lower limb ischemia.
7. Non-atherosclerotic lesion (e.g. vasculitis, dysplasia).
8. Necessary concurrent non-target lesion interventions involving a re-entry device, atherectomy, laser, or ablation procedures, the use of a drug eluting stent, or treatment with any other drug coated balloon.
9. Massive calcifications of the treated lesion (defined as angiographic evidence of dense calcification present on both sides of the vessel wall on two orthogonal views and that extends >50 continuous mm in length; reflective 3 or 4 on the PACSS scale https://doi.org/10.1002%2Fccd.25387).
10. Angiographically confirmed presence of a thrombus in the target lesion.
11. The target lesion requiring primary stenting.
12. Presence of perforation, dissection (Type D or worse) or other injury in target vessel at time of enrollment.
13. Previous bypass graft or stent at target vessel (must be greater than 20mm from target lesion), or iliac stent that cannot permit crossing by the treatment balloon within the introducer sheath Note: In-stent restenosis is not allowed.
14. Gastrointestinal or any other major bleeding in the past three months.
15. Known bleeding disorder or uncontrolled hypercoagulable disorder.
16. Myocardial infarction or any stroke within 30 days prior to the procedure.
17. Known intolerance to required medications (especially antiplatelets and heparin), contrast media (that cannot be adequately pre-medicated), nitinol or paclitaxel.
18. Pregnant and childbearing age women not using effective contraception.
19. Participation in another investigational study (before completing primary endpoint analysis) or previous enrollment to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Safety - MAEs at 12 months | 12 months
  Major Adverse Events (MAEs) at 12 months defined as the composite of: target-limb-related death, major amputation of the target limb and, re-intervention of the target limb.
Efficacy-PAK DCB Success at 12 months, defined as primary patency (PP) | 12 months
  PAK DCB Success at 12 months, defined as primary patency (PP) in the absence of clinically driven bail-out stenting (CDBOS), as defined below.
  Subjects with no CDBOS will be assessed for PP for the purposes of determining True DCB Success. Clinically Driven Bail-Out Stenting (CDBOS): Stents are considered clinically driven when the angiographic core lab determines that a stent was placed after DCB use during the index procedure under the following conditions that were not resolved by prolonged balloon inflation: •Unresolved flow limiting dissection (Type E or F), OR •Residual lumen diameter stenosis > 50% A subject with a CDBOS fails the True DCB success endpoint regardless of patency outcomes.
Primary Patency: Subjects who will achieve primary patency by a combination of duplex ultrasound review and no evidence of clinically driven target lesion revascularization (CD-TLR) prior to the study required 12-month DUS as defined below: | 12 Month
  Duplex Ultrasound Review: A patent target lesion shows a Peak Systolic Velocity Ratio (PSVR) less than 2.5 by the Duplex Ultrasound DUS core lab or Clinically Driven Target Lesion Revascularization CD-TLR: any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed that was considered clinically driven when both of the following conditions were met: Worsening clinical based on an ankle-brachial index (ABI) decrease≥20%or>0.15 compared to maximum early postprocedure ABI or documented increase in Rutherford by at least one class if ABI change was unattainable. Angiographic core lab adjudication of the revascularization angiogram confirming that the target lesion prior to re-intervention demonstrated diameter stenosis >50%.

SECONDARY OUTCOMES:
Technical success rate. | During procedure
  Technical success rate defined as successful balloon insertion, balloon inflation and removal.
Device success defined. | During procedure
  Device success defined as ability to achieve optimal percutaneoustransluminal angioplasty (PTA) outcome (≤30% residual diameter stenosis in post-procedural angiography with no flow-limiting dissection at the target lesion).
Procedural success. | Up to 3 days after index procedure
  Procedural success defined as device success with no major complications. (death, myocardial infarction, amputation, stroke).
Rate of CDBOS. | Up to 3 days after index procedure
  Rate of Clinically Driven Bail-Out Stenting
Primary Patency at 12 months. | 12 months
  Primary Patency at 12 months, defined as target lesion restenosis as determined by DUS (PSVR < 2.5) and freedom from CD-TLR.
Secondary Patency at 12 months. | 12 months
  Secondary Patency at 12 months defined by a PSVR less than 2.5 on DUS regardless of the need for TLR.
Freedom from clinically driven TLR at 30-day follow-up. | 30 days
Freedom from clinically driven TLR at 6-month follow-up. | 6 months
Freedom from clinically driven TLR at 12-month follow-up. | 12 months
Freedom from TVR at 30-day follow-up. | 30 days
Freedom from TVR at 6-month follow-up. | 6 months
Freedom from TVR at 12-month follow-up. | 12 months
All-cause mortality at 30-day follow-up. | 30 days
All-cause mortality at 6-month follow-up. | 6 months
All-cause mortality at 12-month follow-up. | 12 months
Major amputation rate at 30-day follow-up. | 30 days
Major amputation rate at 6-month follow-up. | 6 months
Major amputation rate at 12-month follow-up. | 12 months
Clinical improvement at 30-day follow-up. | 30 days
  Clinical improvement at 30-day follow-up compared to the baseline, defined by Rutherford classification improved by at least one category if ABI improved by at least 20% or 0.15.
Clinical improvement at 6-month follow-up. | 6 months
  Clinical improvement at 6-month follow-up compared to the baseline, defined by Rutherford classification improved by at least one category if ABI improved by at least 20% or 0.15.
Clinical improvement at 12-month follow-up. | 12 months
  Clinical improvement at 12-month follow-up compared to the baseline, defined by Rutherford classification improved by at least one category if ABI improved by at least 20% or 0.15.

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (2):
  - Department of Vascular Surgery; Malopolska Cardiovascular Center; Polish-American Heart Clinics, Chrzanów, Malopolska
  - University Hospital Clinical Hospital No. 2 PUM in Szczecin, Department of General, Dental and Interventional Radiology, Szczecin, West Pomeranian Voivodeship
- Vascular Surgery Teaching Unit CardioVascular Institute Hospital Clinic University of Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buszman PP, Nowakowski P, Milewski K, Orlik B, Zurakowski A, Ludyga T, Polczyk F, Debinski M, Jelonek M, Kachel M, Gasior M, Granada JF, Kiesz RS, Buszman PE. Clinical Randomized Trial Evaluating Novel, Microcrystalline, and Biocompatible Polymer Paclitaxel-Coated Balloon for the Treatment of Femoropopliteal Occlusive Disease: The BIOPAC Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2436-2438. doi: 10.1016/j.jcin.2018.07.029. No abstract available. PMID 30522679